CLINICAL TRIAL: NCT01240551
Title: A Pilot Study of F-18 Sodium Fluoride PET/CT for Metastatic Burden Qualification in Prostate Cancer
Brief Title: F-18 Sodium Fluoride in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Karen Kurdziel, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 110021; 11-C-0021
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Results first posted 2014-12-24 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Prostate Neoplasm
Keywords: Imaging; Bone Metastasis; Bone Scan; Radiopharmaceutical; Pet Scan; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mets via NaF-18 PET/CT (Active Comparator): Patients with known bone metastases (i.e. mets).
  Interventions: Drug: F-18 NaF
- No-Mets via NaF-18 PET/CT (Active Comparator): Patients with no clinical evidence of bone metastases
  Interventions: Drug: F-18 NaF

INTERVENTIONS:
Drug: F-18 NaF — All participants will undergo a static F-18 NaF PET/CT imaging session at baseline, at 4-8 months, and at 10-14 months following enrollment (3 sessions over 1-year). Half of the participants (15 in each group) will undergo two baseline F-18 NaF PET/CT imaging sessions (within 14-days of each other) in order to evaluate the reproducibility of F-18 NaF PET imaging for a total of 4 sessions over a 1-year period.

SUMMARY:
Background:

- Sodium fluoride (NaF) is a common compound that is found in various foods and can be used to increase bone strength. When this compound is added to a small dose of radiation (F-18), it collects in the bones, with higher amounts in areas where the bone is rapidly changing, such as the site of a healing fracture or a tumor. By giving F-18 NaF before a combined positron emission tomography/ computed tomography (PET/CT) scan, researchers hope to be able to better measure the changes in the bone that may indicate that a certain type of cancer (such as prostate cancer) has spread to the bones.

Objectives:

* To evaluate the effectiveness of F-18 NaF in imaging studies to measure bone tumors and their change over time and compare with clinical course, in individuals with prostate cancer.
* To determine the smallest amount of change in the bone tumors that F-18 NaF can accurately measure.

Eligibility:

- Men at least 18 years of age who have been diagnosed with prostate cancer and have had imaging studies to determine whether the cancer has spread to their bones. Both patients with and without known bone involvement will be enrolled.

Design:

* Participants will be screened with a physical examination, medical history, and imaging studies, and will provide baseline blood samples to evaluate kidney function.
* For the study, participants will have two F-18 NaF PET/CT scans on separate days for baseline. These repeat scans will be used to determine the amount of change that is due to the imaging process alone (i.e. not due to the disease getting better or worse. Participants will receive a dose of F-18 NaF intravenously, and will have PET/CT scanning over the body (mid ear to upper thighs) over 1 hour, the body followed by a complete whole-body PET/CT scan at approximately 2 hours after F-18 NaF injection. Participants will be watched closely for side effects from the F-18 NaF until the scans are done, and will be asked to drink plenty of water to void the F-18 NaF from the body after the scans.
* As a followup study, participants will have two more F-18 NaF PET/CT scans, one 4 to 8 months after the first scans and then one 10 to 14 months after the first scans. Participants will provide additional blood samples before the followup scans.

DETAILED DESCRIPTION:
Background:

* Evaluating response to therapy in prostate cancer is limited by the inability to quantify bony metastatic disease
* F-18 sodium fluoride (NaF) is a PET radiopharmaceutical which localizes in regions of bony turnover, and was the 1st bone scan agents (prior to Tc-99m MDP (methylene diphosphonate) availability)
* Today s high sensitivity PET cameras can image the distribution of F-18 NaF as a whole body volume and permit quantification of uptake over time. The addition of co-registered CT increases the diagnostic accuracy for detection of metastatic disease

Primary Objective:

-To evaluate the feasibility of using NaF PET/CT to quantitatively measure the extent of bony metastatic disease in patients with prostate cancer in patients

* To determine the intra-patient reproducibility of F-18 NaF PET/CT
* To explore the relationship between the biodistribution changes in F-18 NaF PET/CT parameters and the clinical response

Eligibility:

* Participant must have pathology proven adenocarcinoma of the prostate.
* Participant must have

  * A history of PSA > 10ng/mL or a history of PSA doubling time of less than or equal to 6 months, and no known bone metastatic involvement on standard of care imaging (Tc-99m MDP bone scan, CT etc).

OR

--Any PSA (prostate specific antigen) level and known bone metastatic disease on standard of care imaging (Tc-99m MDP bone scan, CT etc.)

* Participant must be 18 years or older and have ECOG (Eastern Cooperative Oncology Group) Performance grade of 0 to 2
* Ability to provide informed consent. All subjects must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed.

Design:

This is a pilot, 2-arm, open label study of patients with prostate cancer. One arm will accrue patients with known bone metastases and the second will accrue patient at risk of developing bone metastases (30 patients per group; total enrollment 60 patients). As it is possible that there will be different rates of bone lesion detection dependent on hormone responsiveness of the tumors, further stratification (castrate sensitive vs. castrate resistant tumor) may be performed to evaluate for predominant trends. All participants will undergo a static F-18 NaF imaging session at baseline, at 4-8 months, and at 10-14 months following enrollment (3 sessions over 1-year). Half of the participants (15 in each group) will undergo two baseline F-18 NaF PET/CT imaging sessions (within 14-days of each other) in order to evaluate the reproducibility of F-18 NaF PET imaging for a total of 4 sessions over a 1-year period. The change in bone uptake of F-18 NaF will be measured, reproducibility determined, and preliminary comparisons with clinical response will be made.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants must have a clinical course consistent with prostate cancer and have available documentation of prostate adenocarcinoma from either the National Cancer Institute (NCI) or from an outside pathology laboratory.

Participant must have:

- A history of PSA of > 10ng/mL or a history of PSA doubling time of less than or equal to 6 months, and no known bone metastatic involvement on standard of care imaging (Tc-99m MDP bone scan, CT etc)

OR

- Any PSA level and known bone metastatic disease on standard of care imaging (Tc-99m MDP bone scan, CT etc).

Ability to provide informed consent. All subjects must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed.

EXCLUSION CRITERIA:

Participants with severe claustrophobia unresponsive to oral anxiolytics.

Subjects weighing greater than 350 lbs (weight limit for scanner table), or unable to fit within the imaging gantry.

Subjects with any medical condition or other circumstances that, in the opinion of the Investigator, would significantly decrease obtaining reliable data, achieving study objectives or completing the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-11-30 (Actual); Primary Completion 2013-05-31 (Actual); Study Completion 2013-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen A Kurdziel, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized patient images and associated Prostate Specific-Antigen (PSA) and Gleason Scores.
Time Frame: Indeterminate. Following completion of data analysis de-identified images, PSA and Gleason Scores will be made available on the Cancer Imaging Program's "The Cancer Imaging Archive (TCIA)".
Access Criteria: Open to public.
URL: https://wiki.nci.nih.gov/pages/viewpage.action?pageId=39291472

REFERENCES:
- [Background] Scher HI, Halabi S, Tannock I, Morris M, Sternberg CN, Carducci MA, Eisenberger MA, Higano C, Bubley GJ, Dreicer R, Petrylak D, Kantoff P, Basch E, Kelly WK, Figg WD, Small EJ, Beer TM, Wilding G, Martin A, Hussain M; Prostate Cancer Clinical Trials Working Group. Design and end points of clinical trials for patients with progressive prostate cancer and castrate levels of testosterone: recommendations of the Prostate Cancer Clinical Trials Working Group. J Clin Oncol. 2008 Mar 1;26(7):1148-59. doi: 10.1200/JCO.2007.12.4487. PMID 18309951
- [Background] Tannock IF, de Wit R, Berry WR, Horti J, Pluzanska A, Chi KN, Oudard S, Theodore C, James ND, Turesson I, Rosenthal MA, Eisenberger MA; TAX 327 Investigators. Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1502-12. doi: 10.1056/NEJMoa040720. PMID 15470213
- [Background] Grant FD, Fahey FH, Packard AB, Davis RT, Alavi A, Treves ST. Skeletal PET with 18F-fluoride: applying new technology to an old tracer. J Nucl Med. 2008 Jan;49(1):68-78. doi: 10.2967/jnumed.106.037200. Epub 2007 Dec 12. PMID 18077529
- [Result] Kurdziel KA, Shih JH, Apolo AB, Lindenberg L, Mena E, McKinney YY, Adler SS, Turkbey B, Dahut W, Gulley JL, Madan RA, Landgren O, Choyke PL. The kinetics and reproducibility of 18F-sodium fluoride for oncology using current PET camera technology. J Nucl Med. 2012 Aug;53(8):1175-84. doi: 10.2967/jnumed.111.100883. Epub 2012 Jun 22. PMID 22728263
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0021.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mets Via NaF-18 PET/CT | No-Mets Via NaF-18 PET/CT
Started | 30 | 30
Completed | 26 | 27
Not Completed | 4 | 3
Not completed — Refused further treatment | 3 | 2
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mets Via NaF-18 PET/CT | No-Mets Via NaF-18 PET/CT | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (7.45) | 65.8 (8.67) | 64.98 (8.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 30 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 29 | 30 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 6 | 14
  White | 22 | 24 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Present or Not Present Bone Metastasis
Description: Present and not present bone metastasis was determined by sodium fluoride (NaF) PET (positron emission imaging)/CT (computed tomography) imaging. Present bone metastasis is defined as greater than normal bone uptake. Not present bone metastasis is defined as physiological bone uptake of F-18 NaF on PET/CT imaging (i.e. excluding traumatic and degenerative foci of increased F-18 NaF uptake.
Time Frame: Single imaging sessions will be acquired at baseline, between 4-6 months and between 10-12 months on emolument.
Population: Patient with known prostate cancer. One group with known metastatic bone disease, based on prior clinical imaging scan (Tc-99m bone scan or NaF-18 bone scan or CT, and a second group with clinical risk factors for obtaining bony metastatic disease (i.e. pelvic soft tissue mets, high PSA (prostate specific antigen) blood levels).
Measure: Count of Participants; unit: Participants
Arm/Group | Mets Via NaF-18 PET/CT | No-Mets Via NaF-18 PET/CT
Number analyzed (Participants) | 30 | 30
Participants
  Baseline: Metastasis Present | 30 | 10
  Baseline: Metastasis Not Present | 0 | 20
  4-6 months: Metastasis Present | 29 | 9
  4-6 months: Metastasis not Present | 0 | 20
  10-12 months: Metastasis Present | 26 | 7
  10-12 months: Metastasis Not Present | 7 | 13

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events, see the adverse event module.
Time Frame: date treatment consent signed to date off study, approximately 52.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mets Via NaF-18 PET/CT | No-Mets Via NaF-18 PET/CT
Number analyzed (Participants) | 30 | 30
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 52.5 months.
Description: Adverse events reported were determined NOT to be due to the experimental imaging agent or image, rather the patient disease and/or treatments received.
Arm/Group | Mets Via NaF-18 PET/CT | No-Mets Via NaF-18 PET/CT
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/30 | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mets Via NaF-18 PET/CT (N=30) | No-Mets Via NaF-18 PET/CT (N=30)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0
Renal calculi (Renal and urinary disorders) | 1 (1) | 0
Syncope (Nervous system disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mets Via NaF-18 PET/CT (N=30) | No-Mets Via NaF-18 PET/CT (N=30)
Hematuria (Renal and urinary disorders) | 1 (1) | 0
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0
Pain (General disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No